CLINICAL TRIAL: NCT02798900
Title: The Effect of a Functional Task-training Program Combined With Therapeutic Ultrasound on Pain, Strength, Gait Biomechanics and Functionality in Adults With Hip Osteoarthritis
Brief Title: The Effect of Functional Task Training Combined With Therapeutic Ultrasound on Adults With Hip Osteoarthritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not get funding to develop the clinical trial.
Sponsor: Universidad del Rosario (Other)
Collaborators: CORPORACION HOSPITALARIA JUAN CIUDAD, MEDERI (Unknown)
Responsible Party: Principal Investigator, ROSY PAOLA CARDENAS SANDOVAL, Assistant Professor, Universidad del Rosario
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAP1388
Record Dates: First submitted 2016-05-23; First posted 2016-06-14 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Hip
Keywords: Task-specific exercise; Ultrasonic Waves; Biomechanics; Gait; Rehabilitation; Exercise therapy
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Functional task-training and Ultrasound (Experimental): This group will receive 16 sessions of functional task-training program and therapeutic ultrasound will be applied prior to functional task-training.
  Interventions: Other: Functional task-training; Device: Therapeutic Ultrasound
- Functional task-training (Active Comparator): This group will receive 16 sessions of functional task-training program.
  Interventions: Other: Functional task-training

INTERVENTIONS:
Other: Functional task-training — The functional task-training program includes warming up followed by a functional circuit with muscle strengthening exercises for the major groups of hip oriented to daily life activities and ends with stretching.
Device: Therapeutic Ultrasound — Therapeutic pulsed ultrasound will be applied prior to functional task-training with an intensity of 2.2 W/cm2, frequency of 1 MHz and application time of 4 minutes on the anterior, medial and lateral hip area.
  Arms: Functional task-training and Ultrasound

SUMMARY:
The aim of this study is to evaluate the effect of a functional task-training program combined with therapeutic ultrasound on pain, strength, gait biomechanics and functionality in adults with hip osteoarthritis.

DETAILED DESCRIPTION:
Design

The investigators propose a randomized double blind controlled clinical trial. It would include two comparison groups each with 25 participants with medical diagnosis of hip osteoarthritis classified severity II and III and inclusion criteria of the American College of Rheumatology for the classification and reporting of osteoarthritis of the hip.

All qualified participants will attend a pre-training (baseline) data collection session. During the data collection session, each participant will complete the Western Ontario and MacMaster Osteoarthritis Index (WOMAC). All participants will perform visual analog scale and six minutes walk test for assessing pain and functionality, respectively. They will be assessed their hip muscle strength using manual muscle dynamometer. Their biomechanics gait will be assessed through using an infrared motion capture system, force platforms and motion analysis software (120 Hz, BTS Smart DX100, Italy). All participants in both groups will be asked not to alter their regular physical activity or pain medications during the 15-sessions training program.

Each participant will be assessed pain, strength, gait biomechanics and functionality before and after 16 sessions of intervention. Pain and functionality will be further evaluated in sessions 5th and 10th. The first group will receive 16 sessions of a functional task training program and therapeutic ultrasound versus the second group who will only receive 16 sessions of the same functional task-training program.

Functional task-training program includes warm up, followed by a functional circuit with muscle strengthening exercises for the major groups of hip oriented to daily life activities and ends with stretching. Therapeutic ultrasound will be applied prior to functional task-training with an intensity of 2.2 W/cm2, frequency of 1 MHz and application time of 4 minutes. Temporal average intensity area corresponds to 0.44 W/cm2, the treatment area will be equal to 2 times the effective radiating area on the anterior, medial and lateral hip area.

The hypothesis of this study is the functional-task training program combined with therapeutic ultrasound will decrease the pain, improve the muscle hip strength the gait biomechanics and the functionality of the people with hip osteoarthritis.

In the statistical analysis of the results, the differences will be assessed in the three pain and functionality assessments with a repeated measures using ANOVA; the differences between initial and final measurement of strength, biomechanical gait variables and functionality will be evaluated with a paired Student t-test and Wilcoxon. The differences between groups will be assessed with a t-test for independent samples. Significant differences in the outcomes will be adjusted for covariates with binomial regressions, considering a significance level of p <0.05.

For patient registries:

The Mederi Hospital has an integrated system for collecting, storing, monitoring, reviewing, and reporting on registry data of the participants of the study. It also has a Manual documentation of procedures for each registry, includes protocols and data collection instrument. The manual explains how the investigators should create or assign the patient identification numbers and how duplicate records should be prevented and how to report adverse events.

The hospital takes plans for monitoring or auditing the screening practices trough the auditing department and training to educate data collectors.

Additionally, the investigators will make a Pilot Testing to assess understanding, acceptance and feasibility the patient registry processes.

In the other hand, all staffs involved in data collection will be identified, and their roles and job will be described in data collection and processing.

All data collection will be registered in the integrated system of the Mederi Hospital. The gait biomechanics data will be recorded first in the database of the Smart DX100 system of the Laboratory of Biomechanics if the University of Rosario. The investigators will have an external research (Fulbright Scholar) that will audit the register of the biomechanics data. Then, every participant of the study will have an electronic medical record (EMR) of health-related information.

The Mederi Hospital has a system security plan that includes the policies, standard operating procedures, administrative procedures, electronic signatures and it also has a technical security support.

The plan for missing data where variables are reported as missing,unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results the investigators will quantify the extent of missingness, identifying which individuals have missing data and at which assessment then, the investigators will treat the missing data across a statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hip osteoarthritis

Exclusion Criteria:

* Musculoskeletal disability in other lower extremity joints or trunk
* Acute injuries of lower extremity and trunk in past three months
* Arthroscopic surgery
* An intra-articular injection in past three months
* Candidate for surgery
* Patients with fibromyalgia
* Patients with neurologic disease
* Participation in a structured physical activity program in past three months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for pain | within the first 2 weeks before the intervention
  To measure the pain intensity
Change from Baseline Visual Analog Scale for pain at 16th session of intervention | within the first 2 weeks after the intervention
Muscle strength | within the first 2 weeks before the intervention
  It is the muscle strength of gluteus maximus, medium, quadriceps and hamstrings measured using a manual muscle dynamometer.
Change from Baseline Muscle strength at 16th session of intervention | within the first 2 weeks after the intervention
  Change of the muscle strength of gluteus maximus, medium, quadriceps and hamstrings after the intervention.
Gait biomechanics | within the first 2 weeks before the intervention
  Assess the speed, hip range of motion, and peak hip flexion/extension in the gait phases by using motion analysis system BTS SmartDX100 Brand.
Change from Baseline Gait biomechanics at 16th session of intervention | within the first 2 weeks after the intervention
Six minute walk test (To measure the physical function in terms of the basic mobility) | within the first 2 weeks before the intervention
Change from Baseline Six minute walk test at 16th session of intervention | within the first 2 weeks after the intervention

SECONDARY OUTCOMES:
Change from Baseline Visual Analog Scale for pain at 5th session of intervention | After finishing the 5th session of intervention
Change from Baseline Visual Analog Scale for pain at 10th session of intervention | After finishing the 10th session of intervention
Change from Baseline Six minute walk test at 5th session of intervention | After finishing the 5th session of intervention
Change from Baseline Six minute walk test at 10th session of intervention | After finishing the 10th session of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Songning Zhang, PhD, Study Director — Director, Biomechanics/Sports Medicine Lab, Department of Kinesiology, Recreation, & Sport Studies College of Education, Health and Human Sciences. The University of Tennessee
Locations (1):
- Universidad del Rosario, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oakley EM. Application of continuous beam ultrasound at therapeutic levels. Physiotherapy. 1978 Jun;64(6):169-72. No abstract available. PMID 674399
- [Background] Farcic TS, Baldan CS, Cattapan CG, Parizotto NA, Joao SM, Casarotto RA. Treatment time of ultrasound therapy interferes with the organization of collagen fibers in rat tendons. Braz J Phys Ther. 2013 May-Jun;17(3):263-71. doi: 10.1590/s1413-35552012005000090. PMID 23966143
- [Background] CARTER EF Sr, HARRISS RR, PHILLIPS K, ROBINSON LF. Therapeutic application of ultrasound energy; results of broad clinical survey. J Fla Med Assoc (1914). 1956 Oct;43(4):341-6. No abstract available. PMID 13367362
- [Background] Chan AK, Myrer JW, Measom GJ, Draper DO. Temperature changes in human patellar tendon in response to therapeutic ultrasound. J Athl Train. 1998 Apr;33(2):130-5. PMID 16558499
- [Background] Demchak TJ, Stone MB. Effectiveness of clinical ultrasound parameters on changing intramuscular temperature. J Sport Rehabil. 2008 Aug;17(3):220-9. doi: 10.1123/jsr.17.3.220. PMID 18708676
- [Background] Draper DO, Castel JC, Castel D. Rate of temperature increase in human muscle during 1 MHz and 3 MHz continuous ultrasound. J Orthop Sports Phys Ther. 1995 Oct;22(4):142-50. doi: 10.2519/jospt.1995.22.4.142. PMID 8535471
- [Background] Zhou Q, Lau S, Wu D, Shung KK. Piezoelectric films for high frequency ultrasonic transducers in biomedical applications. Prog Mater Sci. 2011 Feb;56(2):139-174. doi: 10.1016/j.pmatsci.2010.09.001. PMID 21720451
- [Background] ter Haar G. Therapeutic applications of ultrasound. Prog Biophys Mol Biol. 2007 Jan-Apr;93(1-3):111-29. doi: 10.1016/j.pbiomolbio.2006.07.005. Epub 2006 Aug 4. PMID 16930682
- [Background] Hangiandreou NJ. AAPM/RSNA physics tutorial for residents. Topics in US: B-mode US: basic concepts and new technology. Radiographics. 2003 Jul-Aug;23(4):1019-33. doi: 10.1148/rg.234035034. PMID 12853678
- [Background] Draper DO, Sunderland S. Examination of the law of grotthus-draper: does ultrasound penetrate subcutaneous fat in humans? J Athl Train. 1993 Fall;28(3):246-50. PMID 16558239
- [Background] Leighton TG. What is ultrasound? Prog Biophys Mol Biol. 2007 Jan-Apr;93(1-3):3-83. doi: 10.1016/j.pbiomolbio.2006.07.026. Epub 2006 Aug 15. PMID 17045633
- [Background] Stewart HF, Abzug JL, Harris GR. Considerations in ultrasound therapy and equipment performance. Phys Ther. 1980 Apr;60(4):424-8. doi: 10.1093/ptj/60.4.424. PMID 7360798
- [Background] Humphrey VF. Ultrasound and matter--physical interactions. Prog Biophys Mol Biol. 2007 Jan-Apr;93(1-3):195-211. doi: 10.1016/j.pbiomolbio.2006.07.024. Epub 2006 Aug 15. PMID 17079004
- [Background] O'Brien WD Jr. Ultrasound-biophysics mechanisms. Prog Biophys Mol Biol. 2007 Jan-Apr;93(1-3):212-55. doi: 10.1016/j.pbiomolbio.2006.07.010. Epub 2006 Aug 8. PMID 16934858
- [Background] Zeni J Jr, Pozzi F, Abujaber S, Miller L. Relationship between physical impairments and movement patterns during gait in patients with end-stage hip osteoarthritis. J Orthop Res. 2015 Mar;33(3):382-9. doi: 10.1002/jor.22772. Epub 2014 Dec 9. PMID 25492583
- [Background] Eitzen I, Fernandes L, Nordsletten L, Risberg MA. Sagittal plane gait characteristics in hip osteoarthritis patients with mild to moderate symptoms compared to healthy controls: a cross-sectional study. BMC Musculoskelet Disord. 2012 Dec 20;13:258. doi: 10.1186/1471-2474-13-258. PMID 23256709
- [Background] Steinhilber B, Haupt G, Miller R, Grau S, Janssen P, Krauss I. Stiffness, pain, and hip muscle strength are factors associated with self-reported physical disability in hip osteoarthritis. J Geriatr Phys Ther. 2014 Jul-Sep;37(3):99-105. doi: 10.1519/JPT.0b013e3182abe7b5. PMID 24406707
- [Background] Baker KG, Robertson VJ, Duck FA. A review of therapeutic ultrasound: biophysical effects. Phys Ther. 2001 Jul;81(7):1351-8. PMID 11444998
- [Background] Nelson AE, Renner JB, Schwartz TA, Kraus VB, Helmick CG, Jordan JM. Differences in multijoint radiographic osteoarthritis phenotypes among African Americans and Caucasians: the Johnston County Osteoarthritis project. Arthritis Rheum. 2011 Dec;63(12):3843-52. doi: 10.1002/art.30610. PMID 22020742
- [Background] Cibulka MT, White DM, Woehrle J, Harris-Hayes M, Enseki K, Fagerson TL, Slover J, Godges JJ. Hip pain and mobility deficits--hip osteoarthritis: clinical practice guidelines linked to the international classification of functioning, disability, and health from the orthopaedic section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2009 Apr;39(4):A1-25. doi: 10.2519/jospt.2009.0301. No abstract available. PMID 19352008
- [Background] Nicolella DP, O'Connor MI, Enoka RM, Boyan BD, Hart DA, Resnick E, Berkley KJ, Sluka KA, Kwoh CK, Tosi LL, Coutts RD, Havill LM, Kohrt WM. Mechanical contributors to sex differences in idiopathic knee osteoarthritis. Biol Sex Differ. 2012 Dec 23;3(1):28. doi: 10.1186/2042-6410-3-28. PMID 23259740
- [Background] Iversen MD. Managing Hip and Knee Osteoarthritis with Exercise: What is the Best Prescription? Ther Adv Musculoskelet Dis. 2010 Oct;2(5):279-90. doi: 10.1177/1759720X10378374. PMID 22870454
- [Background] Pulsatelli L, Addimanda O, Brusi V, Pavloska B, Meliconi R. New findings in osteoarthritis pathogenesis: therapeutic implications. Ther Adv Chronic Dis. 2013 Jan;4(1):23-43. doi: 10.1177/2040622312462734. PMID 23342245
- [Background] Loeser RF. Age-related changes in the musculoskeletal system and the development of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):371-86. doi: 10.1016/j.cger.2010.03.002. PMID 20699160
- [Background] Bennell KL, Hinman RS. A review of the clinical evidence for exercise in osteoarthritis of the hip and knee. J Sci Med Sport. 2011 Jan;14(1):4-9. doi: 10.1016/j.jsams.2010.08.002. Epub 2010 Sep 17. PMID 20851051
- [Background] Loyola-Sanchez A, Richardson J, MacIntyre NJ. Efficacy of ultrasound therapy for the management of knee osteoarthritis: a systematic review with meta-analysis. Osteoarthritis Cartilage. 2010 Sep;18(9):1117-26. doi: 10.1016/j.joca.2010.06.010. Epub 2010 Jul 14. PMID 20637297
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Murphy LB, Helmick CG, Cisternas MG, Yelin EH. Estimating medical costs attributable to osteoarthritis in the US population: comment on the article by Kotlarz et al. Arthritis Rheum. 2010 Aug;62(8):2566-7; author reply 2567-8. doi: 10.1002/art.27514. No abstract available. PMID 20506219
- [Background] Arokoski J. Pain in hip and knee osteoarthritis. Pain Manag. 2014 May;4(3):177-80. doi: 10.2217/pmt.14.12. No abstract available. PMID 24953071
- [Background] Murphy LB, Helmick CG, Schwartz TA, Renner JB, Tudor G, Koch GG, Dragomir AD, Kalsbeek WD, Luta G, Jordan JM. One in four people may develop symptomatic hip osteoarthritis in his or her lifetime. Osteoarthritis Cartilage. 2010 Nov;18(11):1372-9. doi: 10.1016/j.joca.2010.08.005. Epub 2010 Aug 14. PMID 20713163
- [Background] Sartor CD, Watari R, Passaro AC, Picon AP, Hasue RH, Sacco IC. Effects of a combined strengthening, stretching and functional training program versus usual-care on gait biomechanics and foot function for diabetic neuropathy: a randomized controlled trial. BMC Musculoskelet Disord. 2012 Mar 19;13:36. doi: 10.1186/1471-2474-13-36. PMID 22429765
- [Background] Fernandes L, Storheim K, Nordsletten L, Risberg MA. Development of a therapeutic exercise program for patients with osteoarthritis of the hip. Phys Ther. 2010 Apr;90(4):592-601. doi: 10.2522/ptj.20090083. Epub 2010 Feb 25. PMID 20185613
- [Background] Brosseau L, Wells GA, Pugh AG, Smith CA, Rahman P, Alvarez Gallardo IC, Toupin-April K, Loew L, De Angelis G, Cavallo S, Taki J, Marcotte R, Fransen M, Hernandez-Molina G, Kenny GP, Regnaux JP, Lefevre-Colau MM, Brooks S, Laferriere L, McLean L, Longchamp G. Ottawa Panel evidence-based clinical practice guidelines for therapeutic exercise in the management of hip osteoarthritis. Clin Rehabil. 2016 Oct;30(10):935-946. doi: 10.1177/0269215515606198. Epub 2015 Sep 23. PMID 26400851
- [Background] Monaghan B, Grant T, Hing W, Cusack T. Functional exercise after total hip replacement (FEATHER): a randomised control trial. BMC Musculoskelet Disord. 2012 Nov 28;13:237. doi: 10.1186/1471-2474-13-237. PMID 23190932
- [Background] Eitzen I, Fernandes L, Nordsletten L, Risberg MA. No effects of a 12-week supervised exercise therapy program on gait in patients with mild to moderate osteoarthritis: a secondary analysis of a randomized trial. J Negat Results Biomed. 2015 Mar 5;14:5. doi: 10.1186/s12952-015-0023-y. PMID 25886499
- [Background] Monticone M, Ambrosini E, Rocca B, Lorenzon C, Ferrante S, Zatti G. Task-oriented exercises and early full weight-bearing contribute to improving disability after total hip replacement: a randomized controlled trial. Clin Rehabil. 2014 Jul;28(7):658-68. doi: 10.1177/0269215513519342. Epub 2014 Jan 23. PMID 24459172
- [Background] Outermans JC, van Peppen RP, Wittink H, Takken T, Kwakkel G. Effects of a high-intensity task-oriented training on gait performance early after stroke: a pilot study. Clin Rehabil. 2010 Nov;24(11):979-87. doi: 10.1177/0269215509360647. Epub 2010 Aug 18. PMID 20719820
- [Background] Straudi S, Martinuzzi C, Pavarelli C, Sabbagh Charabati A, Benedetti MG, Foti C, Bonato M, Zancato E, Basaglia N. A task-oriented circuit training in multiple sclerosis: a feasibility study. BMC Neurol. 2014 Jun 7;14:124. doi: 10.1186/1471-2377-14-124. PMID 24906545
- [Background] de Vreede PL, Samson MM, van Meeteren NL, Duursma SA, Verhaar HJ. Functional-task exercise versus resistance strength exercise to improve daily function in older women: a randomized, controlled trial. J Am Geriatr Soc. 2005 Jan;53(1):2-10. doi: 10.1111/j.1532-5415.2005.53003.x. PMID 15667369
- [Background] Hoeksma HL, Dekker J, Ronday HK, Heering A, van der Lubbe N, Vel C, Breedveld FC, van den Ende CH. Comparison of manual therapy and exercise therapy in osteoarthritis of the hip: a randomized clinical trial. Arthritis Rheum. 2004 Oct 15;51(5):722-9. doi: 10.1002/art.20685. PMID 15478147
- [Background] Krauss I, Steinhilber B, Haupt G, Miller R, Martus P, Janssen P. Exercise therapy in hip osteoarthritis--a randomized controlled trial. Dtsch Arztebl Int. 2014 Sep 1;111(35-36):592-9. doi: 10.3238/arztebl.2014.0592. PMID 25249361
- [Background] Koybasi M, Borman P, Kocaoglu S, Ceceli E. The effect of additional therapeutic ultrasound in patients with primary hip osteoarthritis: a randomized placebo-controlled study. Clin Rheumatol. 2010 Dec;29(12):1387-94. doi: 10.1007/s10067-010-1468-5. Epub 2010 May 26. PMID 20499122
- [Background] McQuade KJ, de Oliveira AS. Effects of progressive resistance strength training on knee biomechanics during single leg step-up in persons with mild knee osteoarthritis. Clin Biomech (Bristol). 2011 Aug;26(7):741-8. doi: 10.1016/j.clinbiomech.2011.03.006. Epub 2011 Apr 21. PMID 21514018
- Available data/document: Statistical Analysis Plan — https://uredu-my.sharepoint.com/personal/rosy_cardenas_urosario_edu_co/_layouts/15/guestaccess.aspx?guestaccesstoken=QcFnsRtAu0sL3C3BykRoRmzup56%2fKS1U50PYsgfCPaQ%3d&docid=180e16d39085f4beda2f90ff3f40398ad
- Available data/document: Informed Consent Form — https://uredu-my.sharepoint.com/personal/rosy_cardenas_urosario_edu_co/_layouts/15/guestaccess.aspx?guestaccesstoken=22KPPvsG5ChMhU6k%2bwtjMT9u%2b72A2ABD0JwYpY0D7p8%3d&docid=1b012eb2a38df4685b5d63e2429ba5bcf